CLINICAL TRIAL: NCT06278779
Title: Comparative Effectiveness Study of Two Forms of Ketamine for Treatment-Resistant Depression: a Randomised, Rater-blinded Trial
Brief Title: Comparative Effectiveness Study of Two Forms of Ketamine for Treatment-resistant Depression
Acronym: TREK
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: The George Institute (Other)
Collaborators: The University of New South Wales (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: X23-0311
Record Dates: First submitted 2024-01-20; First posted 2024-02-26 (Actual); Last update posted 2025-06-03 (Actual); Status verified 2025-05

CONDITIONS: Treatment Resistant Depression
MeSH Terms: conditions — Depressive Disorder, Treatment-Resistant | interventions — Esketamine

STUDY DESIGN:
Intervention Model Description: Randomized, prospective, parallel group, comparative effectiveness trial.
Who Masked: Outcomes Assessor
Masking Description: Primary outcome raters will be blinded to treatment allocation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Esketamine group (Active Comparator): Dosing of esketamine intranasal spray will be guided by the Spravato® Product Information. This involves a starting dosage of 28 or 56 mg, with dose adjustment up to 84 mg as required to optimise response. Dose adjustments will be based on effectiveness and tolerability to the previous dose. The recommended treatment protocol is twice per week for 4 weeks, then weekly in weeks 5-8, then option of weekly-fortnightly "maintenance" treatment for responders. After week 8, patients may continue treatment as guided by the ketamine clinic psychiatrist.
  Interventions: Drug: Esketamine group
- Racemic ketamine (Active Comparator): Treatment administration will follow standard clinical practice in the recruiting clinic, with a recommendation to follow an evidence-based and established dose-optimising approach, given by injection, twice per week for 4 weeks, then the frequency of further treatments (week 5 - month 6) will be based on the clinical judgement of the ketamine clinic psychiatrist.
  Dosing will be adjusted by the ketamine clinic psychiatrist, based on clinical response, safety and tolerability. The psychiatrist will review the patient before each treatment, over the first 4 weeks, to judge the dose level required.
  Typically, dosing will begin at the standard dose of 0.5 mg/kg and adjusted using an ascending dose titration schedule if the patient has not shown clinical response and if side effects are adequately tolerated.
  .
  Interventions: Drug: Racemic ketamine

INTERVENTIONS:
Drug: Esketamine group — The recommended dosing for Spravato is:
  Weeks 1-4:
  Starting Day 1 dose:
  < 65 years: 56 mg
  ≥ 65 years: 28 mg
  Subsequent doses:
  28 mg (≥ 65 years), 56 mg or 84 mg twice weekly
  Weeks 5-8:
  28 mg (≥ 65 years), 56 mg or 84 mg once weekly
  From Week 9:
  28 mg (≥ 65 years), 56 mg or 84 mg every 2 weeks or once weekly
  Other Names: Spravato®
  Arms: Esketamine group
Drug: Racemic ketamine — Typically, dosing will begin at the standard dose of 0.5 mg/kg and adjusted as needed using an ascending dose titration schedule:
  1. 0.5 mg/kg
  2. 0.6 mg/kg
  3. 0.75 mg/kg
  4. 0.9 mg/kg
  5. Further increments by 0.1-0.2 mg/kg, up to max 1.5 mg/kg
  Arms: Racemic ketamine

SUMMARY:
The goal of this study is to compare the effectiveness of two formulations of ketamine - Spravato® and racemic ketamine - in people with treatment-resistant depression (TRD). The main questions it aims to answer are:

* How the two formulations compare in terms of their effectiveness in treating TRD.
* How the two formulations compare in their acceptability to patients, safety, effects on patient quality of life and function, and cost effectiveness.

Participants will be randomised to receive either Spravato® or racemic ketamine treatment and asked to complete some questionnaires to assess the effects on mood, treatment acceptability, side effects, quality of life and function, and health economic outcomes.

DETAILED DESCRIPTION:
The TREK study is a randomized, prospective, rater blinded (primary outcome raters), parallel group, comparative effectiveness trial of racemic ketamine and Spravato®, comparing their effectiveness, acceptability, safety, effects on quality of life (QOL), function and cost effectiveness after 4 weeks - 6 months of treatment in people with TRD.

Participants will be recruited from clinics/hospitals that are providing racemic ketamine and Spravato® treatment services for TRD. Participants will be referred, treated and followed up as per the clinic's normal clinical practice. Participants who consent to participate in this research study will undergo other processes in addition to the standard treatment procedures provided by their clinic:

* Randomisation to receive racemic ketamine or Spravato®.
* Completion of questionnaires to measure treatment effects on mood, acceptability, safety, quality of life and function and cost effectiveness.

ELIGIBILITY:
Inclusion Criteria:

* Adult with treatment-resistant depression (TRD: not responded adequately to at least two different antidepressants of adequate dose and duration) who has a current depressive episode (DSM 5)
* Assessed and attested by clinic psychiatrist as appropriate to receive either racemic ketamine or Spravato® ketamine treatment for TRD
* Aged ≥18 years
* Written informed consent for research study obtained

Exclusion Criteria:

* Not able to give informed consent
* Any physical or mental condition which, in the opinion of the investigator, could interfere with study participation including outcome assessments
* Patients who require an interpreter/translator for the clinic consent process, due to the infeasibility of obtaining an interpreter for research assessments, including self-rated scales

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 162 (Estimated)
Dates: Start 2024-06-03 (Actual); Primary Completion 2027-04 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Montgomery-Asberg Depression Rating Scale (MADRS) | From week 0 to week 4.
  Change in score on the Montgomery-Asberg Depression Rating Scale (MADRS). The MADRS is sensitive to change, and is commonly used for treatment trials in depression.
  MADRS includes questions on ten symptoms, each of which yields a score of 0 to 6. The total score ranges from 0 to 60. The higher the MADRS score the more severe the depression. Cutoff points are for levels of depression are:
  0 to 6: normal /symptom absent 7 to 19: mild depression 20 to 34: moderate depression 35 to 60: severe depression.

SECONDARY OUTCOMES:
Montgomery-Asberg Depression Rating Scale (MADRS) score | At week 8, month 4 and month 6
  Score on the Montgomery-Asberg Depression Rating Scale (MADRS). The MADRS is sensitive to change, and is commonly used for treatment trials in depression. See outcome 1 for minimum and maximum values, and whether higher scores indicate a better or worse outcome.
Response - Montgomery-Asberg Depression Rating Scale (MADRS) | Weeks 4, 8 and months 4 and 6
  Response (≥50% improvement in MADRS)
Remission - Montgomery-Asberg Depression Rating Scale (MADRS) | Weeks 4, 8 and months 4 and 6
  Remission (MADRS score ≤10)
DASS-21 | Performed weekly from baseline to week 8 inclusive and at 6 month visit.
  Depression, Anxiety and Stress Scale (DASS-21) - will be used to measure psychological distress. It consists of three 7-item subscales, with items scored on a 4-point Likert scale (0-3) and summed to obtain subscale scores.
Clinical Global Impression-Improvement (CGI-I) | Performed weekly from week 1 to week 4 inclusive, then at week 8 and at 6 month visits.
  The Clinical Global Impression - Improvement scale (CGI-I) is used to assess depressive symptom improvement from study baseline. The minimum value is -6 (maximum deterioration) and the maximum value is 6 (ideal improvement).
Clinical Global Impression-Severity (CGI-S) | Performed weekly from baseline to week 4 inclusive, then at week 8 and at 6 month visits.
  The Clinical Global Impression - Severity scale (CGI-S) is used to assess depressive symptom severity. The minimum value is 1 (normal) and the maximum value is 7 (among the most extremely ill patients).
Columbia Suicide Severity Rating Scale (C-SSRS) | Performed weekly from baseline to week 4 inclusive, then at week 8 and at 6 month visits.
  Columbia Suicide Severity Rating Scale (C-SSRS) - short questionnaire that will be used by the clinic teams as a clinical tool to assess suicidality.
Speed of response - Clinical Global Impression-Improvement (CGI-I) | Performed weekly from week 1 to week 4 inclusive, then at week 8 and at 6 month visits.
  Speed of response, assessed by number of treatments required to attain CGI-I score of ≥ 3.
Psychotomimetic symptoms | Through study completion at each treatment visit, up to 6 months
  Assessed via the Ketamine Side Effect Tool (KSET), designed to monitor the acute, cumulative and longer-term safety of ketamine treatment.
Suicide attempts or gestures | During 6-month study period
  Data collected as an Adverse Event of Special Interest
Number of Participants with urinary symptoms, as assessed using the Bladder Pain/ Interstitial Cystitis Symptom Score (BPIC-SS) | Performed at baseline, week 4, week 8 and at 6 month visit.
  Bladder Pain-Interstitial Cystitis Symptom Score (BPIC-SS) - a self-report symptom-based instrument that identifies moderate to severe bladder pain syndrome. Side effects of racemic ketamine/Spravato® include inflammation of the bladder endothelium. From 8 questions about bladder/urination pain, patients can score a minimum of 0 (asymptomatic) and a maximum of 38 (severe symptoms).
Cognitive Failure Questionnaire scores (CFQ) | Performed at baseline, week 4, week 8 and at 6 month visit.
  Cognitive Failures Questionnaire (CFQ) is a self-rated tool to assess subjective impression of cognitive functioning. From 25 questions, patients can score a minimum of 0 (best) and a maximum of 100 (worst).
Ketamine liking/craving score | Performed at baseline, week 4, week 8 and at 6 month visit.
  Ketamine liking/craving score will be used as a measure of ketamine craving/abuse. A visual analogue scale is used, where patients can score a minimum of 0 (strong dislike/no craving) and a maximum of 30 (very strong liking/constant craving).
Number of Participants with urinary symptoms, as assessed using the Ketamine Side Effect Tool (KSET) | Through study completion at each treatment visit, up to 6 months
  Assessed via the Ketamine Side Effect Tool (KSET), designed to monitor the acute, cumulative and longer-term safety of ketamine treatment.
Acceptability Questionnaire | Performed at week 4, week 8 and at 6 month visit.
  An 8-item self-rated instrument to assess the acceptability of healthcare interventions. This evaluates the constructs of affective attitude, effort burden, ethicality, perceived effectiveness, intervention coherence, self-efficacy, opportunity costs and general acceptability. Patients can score a minimum of 8 (very unacceptable) and a maximum of 40(very acceptable).
  "If reporting a score on a scale, please include the minimum and maximum values, and whether higher scores mean a better or worse outcome." Appears that not all high scores are positive so makes it hard to address this issue.
End of Treatment questionnaire | Used at end of the treatment period(s) over the course of the study.
  Collected via case report form. Captures reason for ceasing, switching or re-starting study medication.
Recovering Quality of Life Questionnaire (REQOL-10) | Over 6 month study period
  Recovering Quality of Life, 10-item (REQOL-10) is used to assess the quality of life for people with different mental health conditions. Patients can score a minimum of 0 (poorest quality of life) and a maximum of 40 (highest quality of life).
WHO Disability Assessment Scale (WHODAS-12) | Over 6 month study period
  12-item WHO Disability Assessment Scale (WHODAS-12) is a 12-item self-rated assessment of health and disability. It will be used to assess functionality. Patients can score a minimum of 0 (no disability) and a maximum of 48 (complete disability).
Patient Health Questionnaire-9 (PHQ-9) | Over 6 month study period
  Patient Health Questionnaire-9 (PHQ-9) is a self-report screening tool designed to assess the severity of depressive symptoms in individuals and monitors symptom changes and treatment effects over time. Patients can score a minimum of 0 (no depression) and a maximum of 27 (severe depression).
Assessment of Quality of Life Questionnaire (AQoL-8D) | Over 6 month study period
  Assessment of Quality of Life Questionnaire (AQoL-8D) consists of 35 items covering 8 dimensions: Independent Living, Pain, Senses, Mental Health, Happiness, Coping, Relationships, and Self-worth. It will be used to assess quality of life outcomes and to facilitate the health economics analysis. There is a max patient score of 1 (perfect health) and a minimum score of 0 (deceased) based on weighted utility scores
Resource Use Questionnaire (RUQ) | Over 6 month study period
  The resource use questionnaire (RUQ) collects information regarding the type and number of contacts with the health system including hospitalisations, consultations and medications. The information is then 'scored' by multiplying indicative unit costs by the number of contacts for each service used. The costs per service are summed to calculate a total health sector cost.
  The resource use questionnaire also collects information regarding time missed (absenteeism) and time working at reduced capacity (presenteeism) for paid work and time missed from unpaid work. The number of hours missed and working at reduced capacity from paid work will be valued using an average wage rate. The hours missed from unpaid work will be valued using a shadow cost for the value of leisure time. These costs are summed and combined with health sector costs to calculate societal costs.
Treatment Preference | Assessed once, prior to randomization
  The Treatment Preferences questionnaire is a simple 3 item self-report questionnaire which asks participants to indicate their treatment preference for one of the 2 interventions, if any; their strength of preference (slight, moderate or strong); their reason for preference (Prefer this method of receiving the medication; Had this treatment before and benefitted; Past negative experience with the other treatment; Impression from reports, other people or media; Other (please specify))
Stanford Expectations of Treatment Scale (SETS) | Assessed once, after randomization and before first treatment
  The SETS is a self-report questionnaire that assesses positive and negative treatment expectations with 6 items rated on a 7-point Likert scale from 0 'not agree at all' to 6 'fully agree'; additional questions ask the responder to confirm the treatment they will receive and whether they have received it before as well as whether any specific benefits or harms/negative side effects are expected
Difficulties in Emotion Regulation Scale-16 (DERS-16) | Performed at baseline and week 4
  The DERS-16 is a self-report measure with established internal consistency, reliability and validity that assesses an individual's typical levels of difficulties in emotion regulation. The DERS-16 assesses five aspects of difficulties in emotion regulation: nonacceptance of emotional responses, difficulty engaging in goal-directed behaviour, impulse control difficulties, limited access to emotion regulation strategies, and lack of emotional clarity.
Level of Personality Functioning Scale-Brief Form (LPFS-BF) | Performed at baseline and week 4
  The LPFS-BF is a 12-item self-report questionnaire that provides a first impression of impairments in personality functioning. The LPFS-BF consists of 12 items, clustered into two higher order domains: self-functioning and interpersonal functioning. Validity and sensitivity have been established in a range of samples and languages

CONTACTS AND LOCATIONS:
Overall Officials: Colleen Loo, Principal Investigator — The University of New South Wales
Locations (6):
- Australia (6):
  - Royal Prince Alfred Hospital, Camperdown, New South Wales
  - Black Dog Institute, Randwick, New South Wales
  - Ramsay Clinic Northside, St Leonards, New South Wales
  - Ramsay Clinic Lakeside, Warners Bay, New South Wales
  - Gold Coast University Hospital, Southport, Queensland
  - Ramsay Clinic Albert Road, Melbourne, Victoria